CLINICAL TRIAL: NCT07278414
Title: Developing and Refining an Intervention to Assess and Address Health-Related Social Needs Among Families of Children With Cancer
Brief Title: Assessing and Addressing Health-Related Social Needs Among Families of Children With Cancer
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00138352; 1K12TR004931-01 (NIH); ONC-PED-2501 (Other: Atrium Health); NCI-2025-08622 (Other: National Cancer Institute)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Childhood Cancers; Caregiver Social Support; Caregiver Distress; Social Needs
Keywords: Social Needs; Caregiver Support; Childhood Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers, Community-Based Organizations, and Healthcare Professionals: Caregivers of children undergoing cancer care, representatives of community-based organizations that provide resources for families of children with cancer, and healthcare providers of children undergoing cancer care
  Interventions: Other: Community Enhancing Resources for Childhood cAncer support (CERCA)

INTERVENTIONS:
Other: Community Enhancing Resources for Childhood cAncer support (CERCA) — CERCA is a context-driven, co-designed intervention leveraging community resources to address unmet Health-related Social Needs (HRSN) among families of children with cancer. This study will observe the process of intervention development and assess acceptability and feasibility.

SUMMARY:
The purpose of this study is to design Community Enhancing Resources for Childhood cAncer support (CERCA) and refine intervention procedures to target Health-related Social Needs (HRSN) in families of children with cancer. CERCA will leverage existing community resources and create partnerships that will lead to sustainable outcomes. The hypothesis is that through context-driven co-design and community-engaged research methods, the study team will develop an acceptable intervention to target unmet HRSN in families of children with cancer.

DETAILED DESCRIPTION:
The first goal of this study is to identify unmet health-related social needs (HRSN) faced by families undergoing pediatric cancer care and identify health system and community resources to address these unmet HRSN. The second goal of this study is to conduct a context assessment of the current processes related to HRSN screening and referrals in the pediatric oncology clinic via individual interviews and clinical workflow observations with healthcare professionals and clinical staff in the pediatric oncology clinic.

Participants of this study will include caregivers of children in cancer care, representatives of community-based organizations that provide resources for families of children with cancer, and healthcare professionals. The study involves virtual or in-person interviews and co-design workshops and will not alter the treatment decisions made by the enrolling investigator or management of the participant's health.

ELIGIBILITY:
Inclusion Criteria:

Caregivers of Children with Cancer

* A caregiver of a child (<18 years old) actively receiving treatment or recently completed treatment (within the past 1 year prior to enrollment) for any type of cancer. A caregiver is defined as any individual involved in bringing the child to the clinic or providing care at home, the hospital, or other healthcare setting (e.g., parents, guardians, siblings, etc.).
* Ability to understand IRB-approved information sheet and willingness to provide consent.
* Age ≥ 18 years at the time of consent.
* Ability to understand the English and/or Spanish language.

Community-based Organizations

* Representative of community-based organizations that provide resources for families of children with cancer
* Ability to understand IRB-approved information sheet and willingness to provide consent.
* Age ≥ 18 years at the time of consent.
* Ability to understand English and/or Spanish language.

Healthcare Professionals

* Physicians, advanced practice practitioners, nurses, clinical social workers, medical assistants, clinic patient service representatives, and cancer center administrators at AHWFBC.
* Ability to understand IRB-approved information sheet and willingness to provide consent.
* Age ≥ 18 years at the time of consent.
* Ability to understand English and/or Spanish language.

Exclusion Criteria:

* There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of all races and ethnicities of 18 years of age or more who meet the eligibility criteria are eligible to participate in this study. No participants will be excluded on the basis of their gender, race, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Unmet Health-Related Social Needs (HRSN) | Baseline
  Identification of unmet health-related social needs (HRSN) faced by families undergoing pediatric cancer care and identify health system and community resources to address these unmet HRSN
Processes of HRSN screening and referrals | Approximately 10 months after study initiation
  Context assessment of the current processes related to HRSN screening and referrals in the pediatric oncology clinic via individual interviews and clinical workflow observations with healthcare professionals and clinical staff in the pediatric oncology clinic.

SECONDARY OUTCOMES:
To develop CERCA (Community Enhancing Resources for Childhood cAncer support) | Approximately 15 months after study initiation
  The CERCA intervention will be co-designed with community-based organizations, caregivers, pediatric oncology healthcare professionals, and cancer center administration. These partners will work alongside the research team via three iterative workshops to: 1) refine the conceptual model for CERCA using data from individual interviews, 2) define intervention features, 3) identify context factors based on context assessment interviews/observations and 4) co-design a protocol of the intervention (e.g., content, decisions on design and tailoring of intervention, and materials).

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M Robles, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Qualitative data only